CLINICAL TRIAL: NCT01024413
Title: A Randomized, Controlled Phase III Trial to Evaluate the Efficacy of Elortinib vs Gefitinib in Advanced Non-small-cell Lung Cancer With EGFR Exon 19 or 21 Mutations
Brief Title: Phase III Trial to Evaluate the Elortinib vs Gefitinib in Advanced NSCLC With EGFR Exon 19 or 21 Mutations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Society of Lung Cancer (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Professor, Chinese Society of Lung Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG0901
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Thoracic Neoplasms
Keywords: Thoracic Neoplasms; Molecular Mechanisms of Pharmacological Action; Protein Kinase Inhibitors; Respiratory Tract Diseases; Lung Neoplasms; Erlotinib; Gefitinib; Epidermal growth factor receptor genes
MeSH Terms: conditions — Thoracic Neoplasms; Respiratory Tract Diseases; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erlotinib (Experimental): erlotinib 150 mg oral till disease progression
  Interventions: Drug: erlotinib
- gefitinib (Active Comparator): gefitinib 250mg oral till disease progression.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: erlotinib — study arm.erlotinib 150 mg oral till disease progression
  Other Names: Tarceva
  Arms: erlotinib
Drug: gefitinib — study arm.gefitinib 250 mg oral till disease progression
  Other Names: Iressa
  Arms: gefitinib

SUMMARY:
This is a randomized controlled trial to compare efficacy and safety between erlotinib and gefitinib in advanced NSCLC harboring EGFR exon 19 or 21 mutations.Eligible patients were randomized to receive erlotinib or gefitinib in any line settings.The primary endpoint was progression-free survival (PFS).

DETAILED DESCRIPTION:
Patients with stage IV NSCLC who have EGFR exon 19 or 21 mutations will randomized to received oral erlotinib 150mg or gefitinib 250mg once daily until disease progression or unacceptable toxicity. Method of direct DNA sequencing of tumor tissue is used to analysis EGFR mutation status of exons 18-21. The response will be evaluated by RECIST criteria first month,second month and then repeat every 3 months after the beginning of the treatment weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB (wet) or IV NSCLC.
* Patients with positive EGFR exon19 or exon21 mutation as confirmed by direct sequencing histologically.
* Signing the informed consent form.
* The vital organ functions are tolerant to therapy.
* Have recovered to CTCAE2 grade below from toxicity of previous chemotherapy and radiotherapy
* PS 0-2 scores.
* Functional reserve of bone marrow is adequate, e.g. white blood cell count ≥3.0×109/L, planet count ≥90×109/L, and HB≥80×109/L.
* Serum bilirubin is 2 times less than the upper limit of normal (ULN), ALT and AST are 3 times less than ULN; for liver metastases, ALT and AST need to be 5 times less than ULN; creatinine should be 2 times less than ULN.

Exclusion Criteria:

* Informed consent is not provided.
* Women of pregnancy or breastfeeding.
* Have difficulty in swallowing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | two years

SECONDARY OUTCOMES:
overall survival | three years
Safety events | two years
Pharmacoeconomic | two years
Response rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yi Long, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thatcher N, Chang A, Parikh P, Rodrigues Pereira J, Ciuleanu T, von Pawel J, Thongprasert S, Tan EH, Pemberton K, Archer V, Carroll K. Gefitinib plus best supportive care in previously treated patients with refractory advanced non-small-cell lung cancer: results from a randomised, placebo-controlled, multicentre study (Iressa Survival Evaluation in Lung Cancer). Lancet. 2005 Oct 29-Nov 4;366(9496):1527-37. doi: 10.1016/S0140-6736(05)67625-8. PMID 16257339
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Fukuoka M, Yano S, Giaccone G, Tamura T, Nakagawa K, Douillard JY, Nishiwaki Y, Vansteenkiste J, Kudoh S, Rischin D, Eek R, Horai T, Noda K, Takata I, Smit E, Averbuch S, Macleod A, Feyereislova A, Dong RP, Baselga J. Multi-institutional randomized phase II trial of gefitinib for previously treated patients with advanced non-small-cell lung cancer (The IDEAL 1 Trial) [corrected]. J Clin Oncol. 2003 Jun 15;21(12):2237-46. doi: 10.1200/JCO.2003.10.038. Epub 2003 May 14. PMID 12748244
- [Background] Giaccone G, Herbst RS, Manegold C, Scagliotti G, Rosell R, Miller V, Natale RB, Schiller JH, Von Pawel J, Pluzanska A, Gatzemeier U, Grous J, Ochs JS, Averbuch SD, Wolf MK, Rennie P, Fandi A, Johnson DH. Gefitinib in combination with gemcitabine and cisplatin in advanced non-small-cell lung cancer: a phase III trial--INTACT 1. J Clin Oncol. 2004 Mar 1;22(5):777-84. doi: 10.1200/JCO.2004.08.001. PMID 14990632
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Bell DW, Lynch TJ, Haserlat SM, Harris PL, Okimoto RA, Brannigan BW, Sgroi DC, Muir B, Riemenschneider MJ, Iacona RB, Krebs AD, Johnson DH, Giaccone G, Herbst RS, Manegold C, Fukuoka M, Kris MG, Baselga J, Ochs JS, Haber DA. Epidermal growth factor receptor mutations and gene amplification in non-small-cell lung cancer: molecular analysis of the IDEAL/INTACT gefitinib trials. J Clin Oncol. 2005 Nov 1;23(31):8081-92. doi: 10.1200/JCO.2005.02.7078. Epub 2005 Oct 3. PMID 16204011
- [Background] Mok T, Wu Y-L, Thongprasert S, et al: Phase III, randomised, open-label, first-line study of gefitinib (G) vs carboplatin/paclitaxel (C/P) in clinically selected patients (PTS) with advanced non-small-cell lung cancer (NSCLC) (IPASS). Ann Oncol 19 (S8): viii1- viii4, 2008 (suppl 8)
- [Background] Jackman DM, Yeap BY, Sequist LV, Lindeman N, Holmes AJ, Joshi VA, Bell DW, Huberman MS, Halmos B, Rabin MS, Haber DA, Lynch TJ, Meyerson M, Johnson BE, Janne PA. Exon 19 deletion mutations of epidermal growth factor receptor are associated with prolonged survival in non-small cell lung cancer patients treated with gefitinib or erlotinib. Clin Cancer Res. 2006 Jul 1;12(13):3908-14. doi: 10.1158/1078-0432.CCR-06-0462. PMID 16818686
- [Background] Riely GJ, Pao W, Pham D, Li AR, Rizvi N, Venkatraman ES, Zakowski MF, Kris MG, Ladanyi M, Miller VA. Clinical course of patients with non-small cell lung cancer and epidermal growth factor receptor exon 19 and exon 21 mutations treated with gefitinib or erlotinib. Clin Cancer Res. 2006 Feb 1;12(3 Pt 1):839-44. doi: 10.1158/1078-0432.CCR-05-1846. PMID 16467097
- [Background] Massuti B, Morán T, Porta R, et al: Multicenter prospective trial of customized erlotinib for advanced non-small cell lung cancer (NSCLC) patients (p) with epidermal growth factor receptor (EGFR) mutations: Final results of the Spanish Lung Cancer Group (SLCG) trial. J Clin Oncol 27:15s, 2009 (suppl; abstr 8023)
- [Background] Yang CH, Yu CJ, Shih JY, Chang YC, Hu FC, Tsai MC, Chen KY, Lin ZZ, Huang CJ, Shun CT, Huang CL, Bean J, Cheng AL, Pao W, Yang PC. Specific EGFR mutations predict treatment outcome of stage IIIB/IV patients with chemotherapy-naive non-small-cell lung cancer receiving first-line gefitinib monotherapy. J Clin Oncol. 2008 Jun 1;26(16):2745-53. doi: 10.1200/JCO.2007.15.6695. PMID 18509184
- [Background] Fukuoka M, Wu YL, Thongprasert S, Sunpaweravong P, Leong SS, Sriuranpong V, Chao TY, Nakagawa K, Chu DT, Saijo N, Duffield EL, Rukazenkov Y, Speake G, Jiang H, Armour AA, To KF, Yang JC, Mok TS. Biomarker analyses and final overall survival results from a phase III, randomized, open-label, first-line study of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer in Asia (IPASS). J Clin Oncol. 2011 Jul 20;29(21):2866-74. doi: 10.1200/JCO.2010.33.4235. Epub 2011 Jun 13. PMID 21670455
- [Background] Costa DB, Schumer ST, Tenen DG, Kobayashi S. Differential responses to erlotinib in epidermal growth factor receptor (EGFR)-mutated lung cancers with acquired resistance to gefitinib carrying the L747S or T790M secondary mutations. J Clin Oncol. 2008 Mar 1;26(7):1182-4; author reply 1184-6. doi: 10.1200/JCO.2007.14.9039. No abstract available. PMID 18309959
- [Derived] Yu YF, Luan L, Zhu FF, Dong P, Ma LH, Li LT, Gao L, Lu S. Modelled Economic Analysis for Dacomitinib-A Cost Effectiveness Analysis in Treating Patients With EGFR-Mutation-Positive Non-Small Cell Lung Cancer in China. Front Oncol. 2021 Dec 14;11:564234. doi: 10.3389/fonc.2021.564234. eCollection 2021. PMID 34970476
- [Derived] Zhou Q, Yang JJ, Chen ZH, Zhang XC, Yan HH, Xu CR, Su J, Chen HJ, Tu HY, Zhong WZ, Yang XN, Wu YL. Serial cfDNA assessment of response and resistance to EGFR-TKI for patients with EGFR-L858R mutant lung cancer from a prospective clinical trial. J Hematol Oncol. 2016 Sep 13;9(1):86. doi: 10.1186/s13045-016-0316-8. PMID 27619632